CLINICAL TRIAL: NCT02305784
Title: Chitinase and Cystic Fibrosis Disease Evolution
Brief Title: Kinetics of YKL-40 Protein in Serum of Cystic Fibrosis Patients
Acronym: Kin_YKL_CF
Status: Completed | Type: Observational
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Yves Berthiaume, Executive Director of the clinic and clinical research, Institut de Recherches Cliniques de Montreal
Other Study IDs: Kin_YKL-40_CF
Record Dates: First submitted 2014-11-11; First posted 2014-12-03 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2017-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Pulmonary exacerbation; inflammation; Chitinase; cytokine; Cystic fibrosis related diabetes
MeSH Terms: conditions — Cystic Fibrosis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will take a blood sample at each regular clinic visit (3-4/year-no evidence of exacerbation in the past two weeks) as well as at the beginning and the end of an exacerbation treated with IV antibiotics.
Oversight: Data Monitoring Committee: No

SUMMARY:
YKL-40 is proposed as a biomarker of various inflammatory disease diabetes and lung disease including cystic fibrosis. In those cross-sectional studies, a unique value of YKL-40 is used to correlate with clinical, physiological, or biological determinants of disease severity (like FEV1 for example in lung disease). There is only one longitudinal study that showed a correlation between circulating levels of YKL-40 and the decline of lung function in smokers sampled from the general population. In order to better understand the potential role of YKL-40 in CF pathophysiology, and to determine its potential role as a biomarker of disease evolution, it is essential to proceed with further clinical evaluation. The investigators propose to perform an observational prospective cohort study to determine if variation of YKL-40 concentration over 24 months correlates with the clinical evolution of the patients.

DETAILED DESCRIPTION:
Observational prospective cohort: The primary objective of the study is to determine if variation of YKL-40 concentration (in blood or sputum) over 24 months will correlate with the biological or clinical condition of the patients. For this study, only patients (FEV1 > 30%) positive for Pseudomonas in the past year will be included, while B Cepacia positive patients will be excluded. There are presently 200 patients meeting these inclusion criteria. The investigators choose to limit the study population to patients with Pseudomonas since they are more likely to have FEV1 changes or clinical evolution during the observation period. The investigators expect a high participation rate since the only obligation for the patients is to provide samples at each visit. A blood (for serum and DNA) and sputum samples will be taken at each regular clinic visit (3-4/year-no evidence of exacerbation in the past two weeks) as well as at the beginning and at the end of an exacerbation treated with IV antibiotics. This will also allow the investigators to determine if there is a change in YKL-40 during an exacerbation. The patients will be followed for a period of 24 months. In parallel to the measurement of YKL-40 in blood and airway secretions, other biological parameters will be monitored (see list below) as well as the BMI, lung function (FEV1/FVC), oxygen saturation and heart rate. The investigators will also monitor the glucose metabolism status of the patient (IGT, CFRD) and the number of exacerbations per year as well as any significant changes in the microbiology status of the patients. A pulmonary exacerbation will be defined as an acute exacerbation of pulmonary symptoms that in the opinion of the CF physician is severe enough to require intravenous antibiotics. The proposed sample size, was shown by power calculation, to be sufficient to demonstrate a meaningful changes in YKL-40 (initial-final) given plausible values of the standard deviation of this difference between patients.

ELIGIBILITY:
Inclusion Criteria:

1. man and woman ≥ 18 ans.
2. documented CF diagnostic (sweat test or genotype).
3. FEV1 ≥ 25%
4. Stable: no infection in the last two weeks before the visit.

Exclusion Criteria:

1. Exacerbation with respiratory symptoms with ou without hospitalization in the last two weeks 2. Exacerbation treated with IV antibiotics. 3. Patients with B. Cepacia

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will follow the patients (<18-year-old) for a period of 24 months. In parallel to the measurement of YKL-40 in blood and airway secretions we will monitor other biological parameters (see list below) as well as the BMI, lung function (FEV1/FVC), oxygen saturation and heart rate. We will monitor the glucose metabolism status of the patient (IGT, CFRD) and the number of exacerbations per year as well any significant changes in the microbiology status of the patients. A pulmonary exacerbation will be defined as an acute exacerbation of pulmonary symptoms that in the opinion of the CF physician is severe enough to require intravenous antibiotics.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2015-05; Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Blood concentration of YKL-40 (ng/ml) | at every outpatient regular visit over a period of 24 months
  Trajectory of YKL-40 over time

SECONDARY OUTCOMES:
Change of Blood concentration of YKL-40 (ng/ml) during an exacerbation | At the beginning and at the end of an exacerbation during the 24 months of follow-up
  Variation of YKL-40 during exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Yves Berthiaume, MD, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- CRIMontreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
not possible since the consent form did not include the possibility to share data with other investigators.